CLINICAL TRIAL: NCT03207685
Title: Characterizing Generalized Seizure Detection And Alerting In The Epilepsy Monitoring Unit With The Empatica Embrace Watch And Smartphone-Based Alert System
Brief Title: Generalized Seizure Detection And Alerting In The EMU With The Empatica Embrace Watch And Smartphone-Based Alert System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Empatica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-002
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Epilepsy
Keywords: Epilepsy; Epilepsy Monitoring Unit; EMU; Seizure; Seizure Detection
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All Subjects (Other): This is a single arm study With a device intervention of Additional Seizure Monitoring
  Interventions: Device: Additional Seizure Monitoring

INTERVENTIONS:
Device: Additional Seizure Monitoring — Embrace could offer an additional layer of seizure monitoring

SUMMARY:
To demonstrate safety and effectiveness of the Embrace device in identifying convulsive seizures (CS) and notifying a caregiver during patient hospitalization at an epilepsy monitoring unit (EMU).

DETAILED DESCRIPTION:
To demonstrate safety and effectiveness of the Embrace device in identifying convulsive seizures (CS) and notifying a caregiver during patient hospitalization at an epilepsy monitoring unit (EMU).

Subjects will be fit with an Embrace device upon admittance into the EMU. The Embrace system will be used in conjunction with the EMU standard care practices to monitor the subject during the subject's stay. EMU standard care practices will not be impacted by the Embrace system, but rather the Embrace will be used to supplement the EMU monitoring. The events detected by Embrace will later be compared to the gold standard results of the video EEG.

A convulsive seizure (CS) is defined for the purpose of this study as any seizure with non-facial motor activity involving one or both upper and/or lower extremities that has repetitive motor activity (rhythmic motor movements).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a history of convulsive seizure (as defined above) who are admitted to a hospital for routine vEEG monitoring related to seizures. Patients who are expected to have a convulsive seizure during their monitoring based on interpretation of clinical history.

Exclusion Criteria:

* Patients who are not expected to have their typical convulsive seizure during the course of their hospital admission (i.e. expected reduction due to anti-epileptic drugs during hospital admission).
* Women who are pregnant.
* Patients who are known or suspected to have a history of PNES only.
* Patients with known allergic reactions to nickel or stainless steel
* Infants who were born pre-term and may not have fully developed skin

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Video-EEG to Embrace System | 6 months
  Lower bound of 95% confidence interval of the positive percent agreement (PPA) greater than 70%, as determined in comparison to Video-EEG adjudicated by 3 independent expert reviewers. A majority rules approach is used to identify convulsive seizures.

SECONDARY OUTCOMES:
Alarm System Comparison | 6 months
  Lower bound of 95% confidence interval of the positive percent agreement (PPA) greater than 70%, as determined in comparison to standard alarm system available in EMU.
False Alarm Rate Tolerability | 6 months
  70% of the EMU staff that use the Embrace consider the false alarm rate to be neutral or better in tolerability based on a survey.
Patient Care Improvement Measure | 6 months
  Embrace maintains or improves the level of patient care, as defined by a survey given to the EMU staff.
Embrace System Usability | 6 months
  Usability of the device perceived by the users (Patients and EMU staff).

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind W Picard, Sc.D., Principal Investigator — Empatica, Inc.
Locations (2):
- NYU Langone Medical Center, New York, New York, United States
- Ospedale Pediatrico Bambino Gesù - Department of Neuroscience, Neurology Unit, Roma, Italy